CLINICAL TRIAL: NCT02472548
Title: A Phase I Randomized, Observer-blind, Controlled, Dose Escalation Trial of the Safety and Tolerability of Two Intramuscular Doses of DPX-RSV(A), a Respiratory Syncytial Virus Vaccine Containing Respiratory Syncytial Virus (RSV) SHe Antigen and a Novel Adjuvant DepoVaxTM, or SHe A Antigen Co-administered With Aluminum Hydroxide, or Placebo to Healthy Adults ≥50-64 Years of Age
Brief Title: A Study to Evaluate the Safety and Reactogenicity of DPX-RSV(A), a Respiratory Syncytial Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Principal Investigator, Joanne Langley, Principal Investigator, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CI1204
Record Dates: First submitted 2015-06-05; First posted 2015-06-16 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Respiratory Syncytial Virus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A, DPX-RSV(A) low dose (Step 1) (Experimental)
  Interventions: Biological: DPX-RSV(A)
- Group B, RSV(A)-Alum low dose (Step 1) (Experimental)
  Interventions: Biological: RSV(A)-Alum
- Group D, DPX-RSV(A) high dose (Step 2) (Experimental)
  Interventions: Biological: DPX-RSV(A)
- Group E, RSV(A)-Alum high dose (Step 2) (Experimental)
  Interventions: Biological: RSV(A)-Alum
- Group C & F, Placebo control (Step 1 and 2) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: DPX-RSV(A) — Prophylactic peptide vaccine targeting RSV will be administered intramuscularly.
  Arms: Group A, DPX-RSV(A) low dose (Step 1); Group D, DPX-RSV(A) high dose (Step 2)
Biological: RSV(A)-Alum — Prophylactic peptide vaccine targeting RSV will be administered intramuscularly.
  Arms: Group B, RSV(A)-Alum low dose (Step 1); Group E, RSV(A)-Alum high dose (Step 2)
Other: Placebo — Normal saline (0.9 % sodium chloride) will be administered intramuscularly.
  Arms: Group C & F, Placebo control (Step 1 and 2)

SUMMARY:
Administration of DPX-RSV(A), a Respiratory Syncytial Virus vaccine containing Respiratory Syncytial Virus (RSV) SHe antigen and DepoVaxTM adjuvant to healthy adults ≥50-64 years of age.

DETAILED DESCRIPTION:
This is a phase 1, First in Humans, randomized (2:2:1) observer blind, controlled, dose ranging, multi-arm parallel-group clinical trial in healthy persons 50 to 64 years of age to assess the safety and immunogenicity of two dose levels of a novel vaccine formulation DPX-RSV(A) consisting of a synthetic Respiratory Syncytial Virus SHe antigen combined with a novel adjuvant DepoVaxTM, compared to the antigen combined with the commonly used adjuvant Aluminum hydroxide, and to a saline placebo control.

The study will evaluate two different doses of DPX-RSV(A) and two doses of the RSV SHe antigen with aluminum hydroxide (RSV(A)-Alum), and a placebo control. The study is randomized, controlled, and observer-blinded in order that allocation to treatment is concealed from the investigative team and the participant. The inclusion of comparator groups (a placebo control group and the RSV(A)-Alum) allows for estimation of the attributable risk of adverse events. Since the study vaccines are not identical in appearance, an unblinded study nurse who has no other role in the study will administer the study vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-64 years, inclusive.
* Good general health status, as determined by history and physical examination no greater than 30 days prior to administration of the test article.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of Diary Cards, return for follow-up visits).
* Written informed consent obtained from the participant.
* If female of child-bearing potential and heterosexually active, has practiced adequate contraception for 30 days prior to injection, has a negative pregnancy test on the day of injection, and has agreed to continue adequate contraception until 180 days after injection. (Please refer to the glossary for the definition of child-bearing potential and adequate contraception).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study product within 28 days preceding the dose of study product, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Planned administration/ administration of a vaccine/product not foreseen by the study protocol within the period starting 28 days before injection of a study vaccine and ending 84 days after.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study product or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination. (Laboratory testing for HIV, Hepatitis C and Hepatitis B will be performed during the screening visit).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drug within 6 months prior to the product dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent). Inhaled and topical steroids are allowed.
* Family history of congenital or hereditary immunodeficiency.
* History of or current autoimmune disease.
* History of hypersensitivity to any test article constituent or products used during the course of study procedures.
* Known or suspected hypersensitivity to any ingredient in the formulation or component of the container.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 180 days of study vaccine receipt.
* Any hematological (hemoglobin level, white blood cell [WBC], and platelet count) and biochemical (alanine aminotransferase [ALT], aspartate aminotransferase [AST], blood urea nitrogen [BUN] and creatinine) abnormality as per local laboratory normal values considered clinically significant by the investigator.
* Transient mild laboratory abnormalities may be rescreened and the participant will be deemed eligible if the laboratory repeat test is normal as per local laboratory normal values and investigator assessment.
* Any acute or chronic, clinically significant disease, as determined by physical examination or laboratory screening tests.
* Malignancies within previous 5 years (excluding non-melanic skin cancer) and lymphoproliferative disorders.
* Current alcoholism and/or drug abuse.
* Acute disease and/or fever at the time of Screening ≥ 38°C

  1. Fever is defined as temperature ≥ 38° /100.4°F by any route; the preferred route for recording temperature in this study will be oral.
  2. Participants with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
  3. Participants with acute disease and/ or fever at the time of Screening may be re-screened at a later date.
* Planned move to a location that will prohibit participating in the trial until study end.
* Any other condition that the investigator judges may interfere with study procedures (e.g. drawing blood) or findings (e.g. immune response).

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and reactogenicity of the intramuscular DPX-RSV(A) | Up to 28 Days after first injection.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety of a second dose of the DPX-RSV(A) | 180 days after vaccination.
The immunogenicity of the DPX-RSV(A) as measured by antibodies directed to the SHe antigen | 28 days after one dose of vaccine and 28 days after a the second dose of a two-dose vaccine schedule as measured by antibodies directed to the SHe antigen.
Persistence of the humoral immune response to two doses of the RSV investigational vaccines, as measured by anti-SHe antibodies | From Day 28 to Day 180 after second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Langley, MD, MSc, FRCPC, Principal Investigator — Dalhousie University, IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada